CLINICAL TRIAL: NCT04955158
Title: Impact of Dexmedetomidine Versus Ketamine Soaked Pharyngeal Packing on Postoperative Sore Throat in Functional Endoscopic Sinus Surgery: a Randomized Double Blind Trial
Brief Title: Dexmedetpmidine Versus Ketamine for Postoperative Sore Throat in Sinus Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar Makram Soliman, Lecturer of anesthesia and ICU, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17101486
Record Dates: First submitted 2021-07-01; First posted 2021-07-08 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Sore Throat
MeSH Terms: conditions — Pharyngitis | interventions — Dexmedetomidine; Ketamine; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dexmedetomidine (Experimental): 75 µg dexmedetomidine soaked pharyngeal pack
  Interventions: Drug: Dexmedetomidine
- Ketamine (Experimental): 50 mg ketamine soaked pharyngeal pack
  Interventions: Drug: Ketamine
- Saline placebo (Experimental): 20 ml 0.9% saline soaked pharyngeal pack
  Interventions: Other: saline 0.9%

INTERVENTIONS:
Drug: Dexmedetomidine — 75 µg dexmedetomidine soaked pharyngeal pack (Group D) putted in the posterior pharyngeal wall after induction of anesthesia and ETT.
  Other Names: Precedex
  Arms: Dexmedetomidine
Drug: Ketamine — 50 mg ketamine soaked pharyngeal pack (Group K) putted in the posterior pharyngeal wall after induction of anesthesia and ETT.
  Other Names: ketalar
  Arms: Ketamine
Other: saline 0.9% — 20 ml 0.9% saline soaked pharyngeal pack (Group C) putted in the posterior pharyngeal wall after induction of anesthesia and ETT.
  Other Names: Normal saline
  Arms: Saline placebo

SUMMARY:
The aim of this randomized clinical trial is to evaluate the impact of dexmedetomidine versus ketamine soaked pharyngeal packing on postoperative sore throat in functional endoscopic sinus surgery (FESS).

DETAILED DESCRIPTION:
A written informed consent was taken from the patients.patients will be randomly assigned to three groups of 40 subjects each; dexmedetomidine or ketamine or saline soaked pharyngeal packs were situated under direct vision. Throat packs made of gauze with a length of 20 cm and a width of 10 cm (folded transverse four times) and medications were diluted with 20 ml normal saline. The packings were placed by the surgeon blinded to the study groups.

1-Dexmedetomidine group: 75 µg dexmedetomidine soaked pharyngeal pack (Group D) putted in the posterior pharyngeal wall after induction of anesthesia and & endotracheal tube (ETT).

2-Ketamine group: 50 mg ketamine soaked pharyngeal pack (Group K) putted in the posterior pharyngeal wall after induction of anesthesia and ETT.

3-Control group: 20 ml 0.9% saline soaked pharyngeal pack (Group C) putted in the posterior pharyngeal wall after induction of anesthesia and ETT.

ELIGIBILITY:
Inclusion Criteria:

* Adults of both sex with American Society of Anesthesiologists (ASA) physical status I-II
* Elective functional endoscopic sinus surgery (FESS) with endotracheal intubation.

Exclusion Criteria:

* A history of preoperative sore throat.
* Upper respiratory tract illness
* Potentially difficult airway
* Patients with history of neck, respiratory or digestive tract pathology
* Chronic smokers
* Using steroid within the last 48 hour
* Pregnant women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2021-08-19 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative sore throat (POST) | 24 hour after surgery
  On arrival in the post anesthesia care unit, the patient was immediately evaluated for the presence of sore throat (time 0 hour) using a standardized scale. The severity of POST was graded on a 4-point scale ranging from 0 to 3; 0 being no sore throat, 1 being mild discomfort (complains only with questioning), 2 being moderate sore throat (complains on their own), and 3 being severe sore throat (change in voice, hoarseness, and throat pain). Evaluations occurred at 0, 1, 2, 4, 6, 12 and 24 hours postoperatively.

SECONDARY OUTCOMES:
Postoperative nausea and vomiting (PONV) score | 2 hours postoperative
  PONV score was assessed and documented using a Verbal Descriptive Scale, which correlates to visual analog nausea scores, with an objective measure of severity: 0 = no PONV: patient reports no nausea and has had no emesis episodes; 1 = mild PONV: patient reports nausea but declines antiemetic treatment; 2 = moderate PONV: patient reports nausea and accepts antiemetic treatment; and 3 = severe PONV: nausea with any emesis episode (retching or vomiting). The score was obtained at 0, 30, 60, 90, and 120 minutes after PACU arrival; 4 mg IV ondansetron for occurred nausea & vomiting.

CONTACTS AND LOCATIONS:
Overall Officials: Omar Soliman, MD, Principal Investigator — Omar makram
Locations (1):
- Omar Soliman, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Higgins PP, Chung F, Mezei G. Postoperative sore throat after ambulatory surgery. Br J Anaesth. 2002 Apr;88(4):582-4. doi: 10.1093/bja/88.4.582. PMID 12066737